CLINICAL TRIAL: NCT04148599
Title: Effect of Intravenous Infusion of Lidocaine in Comparison to Intravenous Infusion of Dexmedetomidine on Proinflammatory Cytokines and Stress Response in Pelviabdominal Cancer Surgeries
Brief Title: Effect of IV Infusion of Lidocaine Compared to IV Infusion of Dexmedetomidine on Proinflammatory Cytokines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Norma Osama Abdalla Zayed (Other)
Collaborators: Abdelhamid, Bassant Mohamed, M.D. (Individual)
Responsible Party: Sponsor-Investigator, Norma Osama Abdalla Zayed, Assistant lecturer of anesthesia, National Cancer Institute, Egypt
Organization: National Cancer Institute, Egypt (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 201617050.3
Record Dates: First submitted 2019-09-24; First posted 2019-11-01 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2019-10

CONDITIONS: Inflammatory Response

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- dexmedetomidine (Active Comparator): dexmedetomidine ( precedex) infusion will be administered preoperatively and continued intraoperatively
  Interventions: Drug: dexmedetomidine infusion
- lidocaine (Active Comparator): Lidocaine (Xylocaine) infusion will be administered preoperatively and continued intraoperatively
  Interventions: Drug: lidocaine infusion
- placebo (Placebo Comparator): saline infusion will be administered preoperatively and continued intraoperatively
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: dexmedetomidine infusion — a loading dose of 1µg/kg of dexmedetomidine (precedex) made to 50 ml using normal saline will be given over 10 minutes followed by infusion of dexmedetomidine with a dose of 0.5µg/kg/hour till the end of surgery.
  Arms: dexmedetomidine
Drug: lidocaine infusion — a loading dose of 1.5 mg/kg of lidocaine made to 50 ml using normal saline and given over 10 minutes followed by infusion of lidocaine with a dose of 1.5 mg/kg/hour till the end of surgery.
  Arms: lidocaine
Drug: Placebos — 50 ml of normal saline given over 10 minutes followed by saline infusion intraoperatively at a rate of 10 ml/hour till the end of surgery.
  Arms: placebo

SUMMARY:
This study is designed to compare between intravenous infusion of dexmedetomidine and intravenous infusion of lidocaine in reduction of proinflammatory cytokines as IL-6 and TNF-α, some stress reactions (serum insulin and serum lactate),and postoperative analgesic requirements in patients undergoing surgery for pelviabdominal cancers.

DETAILED DESCRIPTION:
Cancer patients who undergo surgery face many sources of stress. Surgery causes major cytokine and neuroendocrinal changes like increased levels of catecholamine and steroid hormones and other metabolic consequences .This stress response is considered a defense mechanism important for developing resistance to noxious insults.

The cytokine cascade caused by surgical stimulation is complex with various effects on the injured host. Increased production of proinflammatory cytokines from the site of injury causes many systemic changes such as metabolic derangements and hemodynamic instability. Some released cytokines like tumor necrosis factor alpha (TNF-α) and Interleukin 6(IL-6) can cause long lasting hyperalgesia. These proinflammatory cytokines change pain signal transmission through cytokine induced release of some neuroactive substances like nitric oxide, oxygen free radicals and excitatory amino acids. On the other hand anti-inflammatory cytokines are also released during inflammation to counteract these effects and keep balance.

Dexmedetomidine is a highly selective alpha-2 adrenergic receptor agonist that has sedative, analgesic, anesthetic-sparing properties with no respiratory depression. Its anti-inflammatory effects are being studied.

Intravenous lidocaine can be used in management of chronic pain. Lidocaine has anti-inflammatory properties and is capable of reducing postoperative analgesic requirements and the length of hospitalization.

The effect of both drugs on proinflammatory cytokines and stress response will be assessed

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesia (ASA) Physical Status classification:

ASA II physical status.

* Age between 18 to 60 years old.
* Patients who will undergo major pelviabdominal surgery.

Exclusion Criteria:

* Patient refusal.
* Allergy to local anesthetics.
* Cognitive disorders.
* uncontrolled diabetes or hypertension.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-06-13 (Actual)

PRIMARY OUTCOMES:
change in inflammatory mediators | preoperative (baseline), immediately postoperative and 24 hours postoperative
  change in plasma levels of IL-6 (pg/ml), TNF-α (pg/ml)
change in serum level of insulin and lactate | preoperative (baseline), immediately postoperative and 24 hours postoperative
  change in serum levels of insulin (ng/ml) and lactate (ng/ml)

SECONDARY OUTCOMES:
Rescue analgesia | 1st 24 hours
  time of first rescue analgesia
Visual analogue scale (VAS) score for pain | at 0 hour, 2 hour,6 hour, 12 hour and 24 hour
  assessment of postoperative pain using the visual analogue scale score. the scale is a straight horizontal line (100 mm). The ends are defined as the extreme limits of pain orientated from the left (no pain) to the right (worst pain).The patient marks on the line the point that they feel represents their perception of their current state.
  The VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patient marks.higher VAS score means worse pain
postoperative morphine requirements | 1st 24 hours
  total morphine consumption (mg)

CONTACTS AND LOCATIONS:
Overall Officials: Emad Gerges, MD, Study Director — National Cancer Institute (NCI)
Locations (1):
- National cancer institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No